CLINICAL TRIAL: NCT06783270
Title: T-cell Therapy with CRISPR PD1-edited Tumor Infiltrating Lymphocytes for Patients with Metastatic Melanoma
Acronym: CRISPR-TIL
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Inge Marie Svane (Other)
Responsible Party: Sponsor-Investigator, Inge Marie Svane, MD, professor, center leader, Herlev Hospital
Organization: Herlev Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MM2318; 2023-510417-25-01 (EU CTIS Number)
Record Dates: First submitted 2024-12-13; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Melanoma Metastatic
Keywords: TIL-therapy; TIL-ACT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous CRISPR-PD1 modified tumor infiltrating lymphocytes (Experimental): Tumor infiltrating lymphocytes expanded ex vivo from an excised tumor and treated with CRISPR-Cas9 to effectively silence the PD-1 coding gene in the T-cells. This is given as an intravenous infusion after lymphodepleting chemotherapy using cyclophosphamide and fludarabine-phosphate and followed by up to 6 doses of high-dose interleukin-2 infusions.
  Interventions: Biological: TIL therapy

INTERVENTIONS:
Biological: TIL therapy — Compared to traditional TIL-therapy, this study will include silencing of the PD-1 coding gene in the TILs using non-viral CRISPR-Cas9 prior to the rapid expansion protocol.

SUMMARY:
The purpose of this study is to assess wether it is safe and feasible to treat patients with tumor infiltrating lymphocytes that have been silenced for PD-1, using CRISPR-Cas9.

DETAILED DESCRIPTION:
In this study the investigators will treat patients with advanced (inoperable) or metastatic melanoma with tumor infiltrating lymphocytes (TILs) in combination with lymphodepleting chemotherapy and high-dose interleukin-2. The TILs are harvested from a patient tumor and expanded a thousand-fold in a laboratory over approximately 6 weeks before being infused back into the patient. This is a well known and tried treatment regimen, often called TIL-therapy or TIL-ACT. In this study the investigators will add CRISPR-Cas9 modification to the production process of the TILs to silence the expression of PD-1 on the surface of the infused cells. The aim of this study is to demonstrate wether treatment with these PD1-deficient TILs (CRISPR-TILs) is safe and feasible.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed inoperable or metastatic melanoma (stage IIIc or IV).
2. Progressive disease after standard treatment with anti-PD-1 check-point inhibition or combination of aforementioned with anti-CTLA-4 check-point inhibition.
3. Age: 18 - 75 years at the time of signed Informed consent.
4. ECOG performance status of ≤1 (Appendix 2).
5. Is fit for tumor resection and has at least one lesion (> 1 cm3) available for surgical resection for manufacture of TIL. (Unless TILs are already available through metastasectomy prior to enrollment in this study, as described in step one under study design)
6. At least one measurable parameter in accordance with RECIST 1.1 -criteria (excluding the lesion to be resected).
7. LVEF assessment with documented LVEF ≥50% by either TTE or MUGA.
8. Sufficient organ function, including:

   * Absolute neutrophil count (ANC) ≥ 1.500 /μl
   * Leucocyte count ≥ lower normal limit
   * Platelets ≥ 100.000 /μl and <700.000 /μl
   * Hemoglobin ≥ 6.0 mmol/l
   * eGFR > 70
   * S-bilirubin ≤ 1.5 times upper normal limit (Exception: Subjects with liver metastasis ≤ 2.5 × ULN)
   * ASAT/ALAT ≤ 2.5 times upper normal limit (Exception: Subjects with liver metastasis ≤ 5.0 × ULN)
   * Alkaline phosphatase ≤ 5 times upper normal limit
   * Lactate dehydrogenase ≤ 5 times the upper normal limit
   * Sufficient coagulation: APPT<40 and INR<1.5
9. Signed statement of consent after receiving oral and written study information
10. Willingness to participate in the planned controls and capable of handling toxicities.
11. Subject must receive CRISPR-TIL as the next therapy following tumor resection unless bridging therapy is administered:

    * Bridging therapy is discouraged. However, if in the opinion of the Investigator, the subject requires immediate therapy after tumor resection, the subject may receive bridging therapy for the period during which the subject is awaiting the manufacture of TIL-infusion product. Bridging therapy may be a continuation of the therapy the subject was receiving prior to tumor resection or may be a new therapy.
    * Following this bridging therapy, the subject must adhere to the mandatory washout periods (described in exclusion criterion 1) and must continue to have measurable disease prior to receiving CRISPR-TIL.
12. Age and Reproductive Status:

    * Women of childbearing potential (WOCBP) must have a negative urine or serum pregnancy test AND must agree to use an effective method of contraception starting at the first dose of chemotherapy for at least 12. WOCB must also agree to refrain from egg donation, storage, or banking during these same time periods. The following are considered safe methods of contraception:

      * Hormonal anticonception (birth control pills, spiral, depot injection with gestagen, subdermal implantation, hormonal vaginal ring, and transdermal depot patch)
      * Intrauterine device
      * Surgical sterilization
      * Surgical sterilization of male partner with verification of no sperm after the procedure
      * Menopause (for more than 12 months)
    * Male subjects must be surgically sterile or agree to use a double-barrier contraception method or abstain from sexual activity with an WOCBP starting at the first dose of chemotherapy and for 6 months thereafter. Male subjects must also agree to refrain from sperm donation, storage, or banking.

Exclusion Criteria:

1. Subject has received or plans to receive the following therapy/treatment prior to tumor resection (TR) or lymphodepleting chemotherapy (LDC):

   * Cytotoxic chemotherapy: Washout period 3 weeks before TR and LDC.
   * Small molecules/TKI: Washout period 1 week before TR and LDC.
   * Immune therapy (monoclonal AB therapy, CPI, and biologics): 2 weeks before TR and LDC
   * Prior T-cell therapy, including gene therapy using an integrating vector.
   * Corticosteroids at dose equivalent > 10 mg prednisone or any other immunosuppressive therapy. 2 weeks before TR and LDC. Note: Use of topical steroids is not an exclusion.
   * Investigational treatment: 4 weeks or 5 half-lives, whichever is shorter before TR and LDC.
   * Radiation to the pelvis and/or multiple bones containing ≥ 25% of bone marrow: 4 weeks before TR and LDC.
   * Whole brain radiotherapy or brain stereotactic radiosurgery: 4 weeks before TR and LDC.
   * Radiotherapy to the target lesions: 3 months prior to TIL infusion. A lesion with unequivocal progression post-radiotherapy may be considered a target lesion.
2. A history of prior malignancies. Patients treated for another malignancy can participate if they are without signs of disease for a minimum of 2 years after treatment. Subjects with curatively treated ductal carcinoma in situ (DCIS or LCIS) breast cancer for which they are taking hormonal therapy is acceptable. Resectable squamous or basal cell carcinoma of the skin is acceptable.
3. Patients with metastatic ocular/mucosal or other non-cutaneous melanoma. Unknown primary melanoma is eligible.
4. Toxicity from previous anti-cancer therapy must have resolved to ≤ Grade 1 or baseline prior to enrollment (except for non-clinically significant toxicities e.g., alopecia, vitiligo). Subjects with Grade 2 toxicities who are deemed stable or irreversible (e.g., peripheral neuropathy) can be enrolled.
5. Patients who have more than 2 CNS metastases or who have any CNS lesion that is symptomatic, greater than 1 cm in diameter, or show significant surrounding edema on MRI scan will not be eligible until they have been treated and demonstrated no clinical or radiologic CNS progression for at least 2 months.
6. The following patients will be excluded because of their inability to receive high-dose interleukin-2 (See appendix 5):

   * History of coronary revascularization
   * Documented LVEF of less than 45% in patients with clinically significant atrial and/or ventricular arrhythmias including but not limited to atrial fibrillation, ventricular tachycardia, 2o or 3o heart block
   * Documented FEV-1 less than or equal to 60% predicted value for patients with: A prolonged history of cigarette smoking (greater than 20 pack years), large tumor burden in the lungs, or Symptoms of respiratory distress.
7. Known hypersensitivity to one of the active drugs or one or more of the excipients.
8. Severe medical conditions, such as severe asthma/COLD, significant cardiac disease, and poorly regulated insulin-dependent diabetes mellitus among others.
9. Creatinine clearance (eGFR) < 70 ml/min*.
10. Acute/chronic infection with HIV, hepatitis, and syphilis among others.
11. Severe allergies or previous anaphylactic reactions.
12. Active autoimmune or immune-mediated disease that has not yet resolved. Subjects with the following will be eligible:

    * Immune-mediated AEs secondary to immunotherapy which have resolved to ≤ Grade 1 without steroids;
    * Hypothyroidism, Type I diabetes, adrenal insufficiency, or pituitary insufficiency that are stable on replacement therapy;
    * Disorders such as asthma, vitiligo, psoriasis, or atopic dermatitis that are well-controlled without requiring systemic immunosuppression;
    * Other stable immune conditions that do not require prednisone higher than 10 mg/day or their equivalent dose for other corticosteroid agents may be acceptable with the agreement of the Sponsor.
13. Pregnant women and women breastfeeding.
14. Subjects deemed unlikely to fully comply with protocol requirements by the study investigator.

    * In selected cases it can be decided to include a patient with a eGFR < 70 ml/min with the use of a reduced dose of chemotherapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-12-16 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | From surgery to CRISPR-TIL infusion (5-10 weeks)
  Assess feasibility measured by the number of subjects who undergo surgery and successfully undergo CRISPR-TIL infusion
Incidence rate of treatment-emergent adverse events | From admission to 2nd evaluation (3 months after CRISPR-TIL infusion)
  Determine the safety and tolerability measured by the incidence rate of grade 3 treatment-emergent adverse events and serious adverse events by severity and their relationship to the CRISPR-TIL infusion.

SECONDARY OUTCOMES:
Objective response rate | From treatment until the 12 months evaluation scan.
  Assess the clinical effect of the treatment by use of the objective response rate (using RECIST 1.1).

CONTACTS AND LOCATIONS:
Locations (1):
- CCIT-DK, Herlev, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No
Due to a small patient cohort, all individual patient data will be recognizable and assignable to the persons themselves

REFERENCES:
- [Background] Chamberlain CA, Bennett EP, Kverneland AH, Svane IM, Donia M, Met O. Highly efficient PD-1-targeted CRISPR-Cas9 for tumor-infiltrating lymphocyte-based adoptive T cell therapy. Mol Ther Oncolytics. 2022 Jan 10;24:417-428. doi: 10.1016/j.omto.2022.01.004. eCollection 2022 Mar 17. PMID 35141398
- See also: CTIS registration — https://euclinicaltrials.eu/search-for-clinical-trials/?lang=en&EUCT=2023-510417-25-01